CLINICAL TRIAL: NCT03739554
Title: A Phase I Combination Study of CYC065 and Venetoclax for Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Brief Title: CYC065 CDK Inhibitor and Venetoclax Study in Relapsed/Refractory CLL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYC065-02
Record Dates: First submitted 2018-10-01; First posted 2018-11-14 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Relapsed or Refractory Chronic Lymphocytic Leukemia
Keywords: CYC065; CDK2/9; venetoclax; BCL-2; MCL-1; Relapsed; Refractory; chronic lymphocytic leukemia; small lymphocytic lymphoma
MeSH Terms: conditions — Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — CYC065; venetoclax

STUDY DESIGN:
Intervention Model Description: Three to 6 patients will be entered at a given CYC065 dose level. Dose escalation will be 33% until one out of 3 patients experienced a DLT at a given dose level. Dose escalation will continue at 25% if no additional DLT is observed; otherwise, dose escalation will be stopped. At least 6 patients will be treated at RD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CYC065 and venetoclax (Experimental): CYC065 will be administered intravenously via 4-hour infusion on Day 1 and Day 15 after the venetoclax ramp-up schedule is completed. Venetoclax will be taken daily at a dose that is deemed safe and tolerable after the ramp-up schedule. One cycle will be 28 days or 4 weeks.
  Interventions: Drug: CYC065; Drug: Venetoclax

INTERVENTIONS:
Drug: CYC065 — intravenous infusion
Drug: Venetoclax — oral capsule
  Other Names: ABT-199

SUMMARY:
A Phase I Combination Study of CYC065 and Venetoclax for Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)

DETAILED DESCRIPTION:
This is an open-label, single arm, dose escalation study in patients with relapsed or refractory CLL. Treatment will be administered on an outpatient basis and all patients will receive CYC065 over 4-hour infusion once every 2 weeks on Day 1 and Day 15 in combination with venetoclax. One treatment cycle is 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* CLL that is relapsed or refractory to BTK inhibitors and is on a stable dose of venetoclax
* ECOG 0-2
* Adequate bone marrow function
* Adequate renal function
* Adequate liver function
* INR <=1.2 in patients not receiving chronic anticoagulation
* At least 4 weeks from prior cytotoxic chemotherapy
* At least 4 weeks from major surgery
* Agree to practice effective contraception

Exclusion Criteria:

* Known CLL involvement in CNS that is symptomatic and active
* currently receiving radiotherapy, biological therapy, or any other investigational agents
* Uncontrolled intercurrent illness
* Pregnant or lactating
* Known to be HIV-positive
* Known active hepatitis B and/or hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Number of patients who experience dose-limiting toxicity (DLT) | At the end of cycle 1 (each cycle is 28 days)

SECONDARY OUTCOMES:
Pharmacokinetic effect | At the end of cycle 1 (each cycle is 28 days)
  Plasma drug level
Pharmacodynamic effect | At the end of cycle 1 (each cycle is 28 days)
  MCL-1 level in peripheral white blood cells

OTHER OUTCOMES:
Anti-tumor activity | From the date of first dose of CYC065 to 4 weeks after the last dose of CYC065
  Response assessed by investigators based on International Workshop for CLL criteria or International Working Group criteria for patients with small lymphocytic lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kirschbaum, MD, Study Director — Cyclacel Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Investigational Site, Baltimore, Maryland
  - Investigational Site, Charlotte, North Carolina
  - Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: No